CLINICAL TRIAL: NCT03364985
Title: A Phase I, Randomized, Double-blind, Placebo- and Active-controlled, Single- and Multiple-ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of DWP16001 Following Oral Administration in Healthy Male Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DWP16001 After Oral Administration in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP16001001
Record Dates: First submitted 2017-11-29; First posted 2017-12-07 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1: DWP16001 Amg (Experimental): DWP16001 Amg, tablets, orally, single dose administration
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 2: DWP16001 Bmg (Experimental): DWP16001 Bmg, tablets, orally, single dose administration
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 3: DWP16001 Cmg (Experimental): DWP16001 Cmg, tablets, orally, single dose administration
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 4: DWP16001 Dmg (Experimental): DWP16001 Dmg, tablets, orally, single dose administration
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 5: DWP16001 Emg (Experimental): DWP16001 Emg, tablets, orally, single dose administration
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 6: DWP16001 Fmg (Experimental): DWP16001 placebo-matching tablets, Active-control placebo-matching tablets, orally, repeated dose administration(for 15days)
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 7: DWP16001 Gmg (Experimental): DWP16001 placebo-matching tablets, Active-control placebo-matching tablets, orally, repeated dose administration(for 15days)
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 8: DWP16001 Hmg (Experimental): DWP16001 placebo-matching tablets, Active-control placebo-matching tablets, orally, repeated dose administration(for 15days)
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 9: DWP16001 Img (Experimental): DWP16001 placebo-matching tablets, Active-control placebo-matching tablets, orally, repeated dose administration(for 15days)
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin
- Cohort 10: DWP16001 Jmg (Experimental): DWP16001 placebo-matching tablets, Active-control placebo-matching tablets, orally, repeated dose administration(for 15days)
  Interventions: Drug: DWP16001; Drug: Placebo; Drug: Dapagliflozin

INTERVENTIONS:
Drug: DWP16001 — DWP16001 tablets
Drug: Placebo — DWP16001 placebo-matching tablets, Active control placebo-matching tablets
Drug: Dapagliflozin — Forxiga®

SUMMARY:
This is a dose block-randomized, double-blind, placebo- and active-controlled, single and multiple dosing, dose-escalation clinical phase 1 trial to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of DWP16001 after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults aged 19 to 50 at the time of screening test.
2. Body weight between 50.0 kg and 90.0 kg and Body Mass Index (BMI) between 18.0 and 27.0.
3. Written consent on voluntary decision of participation prior to the screening procedure after being fully informed of and completely understanding this study.
4. Eligible to participate in the study by discretion of the investigator following medical examination by interview, physical examination, and clinical examination.

Exclusion Criteria:

1. Presence of a clinically significant hepatic, renal, nervous, respiratory, endocrine, blood•tumor, cardiovascular, urogenital, psychiatric disorder or prior history.
2. Presence or prior history of a gastrointestinal disorder (e.g., gastrointestinal ulcers, gastritis, stomach cramps, gastroesophageal reflux disease, Crohn's disease, etc.), or prior history of surgery (except for simple appendectomy or hernia surgery) that may affect safety and PK/PD assessment.
3. Hypersensitivity to a drug containing an ingredient of the investigational product (DWP16001), Dapagliflozin or similar ingredient or other drugs (e.g., aspirin, antibiotics, etc.) or medical history of clinically significant hypersensitivity.
4. Following laboratory abnormalities identified during the screening test:

   * AST (SGOT), ALT (SGPT) >1.5 upper limit of normal range
   * Creatinine clearance calculated by the MDRD equation < 90 mL/min
   * Repeatedly confirmed QTc interval > 450 ms
   * Fasting serum glucose > 110mg/dL or < 70mg/dL
   * Serum HbA1c > 6.5 mg/dL

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2017-12-03 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Number and percentage of Participants With Adverse Events (AE) | Day -2(Randomization) to Day 8~12(Post-study visit) in single ascending dose or Day-3d to Day 22~ (Post-study visit)
  All AE standardized using MedDRA was assessed by investigator using the protocol defined grading system. Intensity was categorized as mild, moderate and severe
Number and percentage of Participants With Adverse Drug Reactions (ADR) | Day -2(Randomization) to Day 8~12(Post-study visit) in single ascending dose or Day-3d to Day 22~ (Post-study visit)
  An adverse drug reaction (ADR) is an injury caused by taking an investigational product
Number of Participants With Clinically Significant Vital Sign findings | Day -2(Randomization) to Day 8~12(Post-study visit) in single ascending dose or Day-3d to Day 22~ (Post-study visit)
  Blood pressure, pulse and body temperature were tested. The Average, Median, Standard Deviation, Min, Max values will be calculated to assess the safety/tolerability
Number of Participants With Clinically Significant Electrocardiogram(12-lead ECG) findings | Day -2(Randomization) to Day 8~12(Post-study visit) in single ascending dose or Day-3d to Day 22~ (Post-study visit)
  Ventricular rate, RR interval, PR interval, QRS duration, QTcB and QTcF were recorded. The results of 12-lead ECG will be categorized Normal/Abnormal NCS(No clinically significant)/Abnormal CS(clinically significant).
Number of Participants With Clinically Significant Laboratory results | Day -2(Randomization) to Day 8~12(Post-study visit) in single ascending dose or Day-3d to Day 22~ (Post-study visit)
  Hematology, Blood chemistry, Coagulation and Urinalysis were tested. The Average, Median, Standard Deviation, Min, Max values will be calculated to assess the safety/tolerability.

SECONDARY OUTCOMES:
Cmax: Maximum concentration of DWP16001 | 0 hour (pre-dose), 0.25 hour, 0.5 hour, 0.75 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 12hour, 24 hour, 36 hour, 48 hour, 72 hour
  in single ascending dose cohort
Cmax,ss: Maximum concentration of DWP16001 at steady state | Day1 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour, Day 4, 7, 10, 13 0 hour (pre dose), Day 15 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in multiple ascending dose cohort
Cmin,ss: Minimum concentration of DWP16001 at steady state | Day1 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour, Day 4, 7, 10, 13 0 hour (pre dose), Day 15 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in multiple ascending dose cohort
Time of maximum concentration | 0 hour (pre-dose), 0.25 hour, 0.5 hour, 0.75 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 12hour, 24 hour, 36 hour, 48 hour, 72 hour
  in single ascending dose cohort
Tmax,ss: Time of maximum concentration at steady state | Day1 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour, Day 4, 7, 10, 13 0 hour (pre dose), Day 15 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in multiple ascending dose cohort
AUClast: Area under the plasma concentration-time curve from time 0 to 72hours | 0 hour (pre-dose), 0.25 hour, 0.5 hour, 0.75 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 12hour, 24 hour, 36 hour, 48 hour, 72 hour
  in single ascending dose cohort
AUCinf: Area under the plasma concentration-time curve from time 0 to infinity | 0 hour (pre-dose), 0.25 hour, 0.5 hour, 0.75 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 12hour, 24 hour, 36 hour, 48 hour, 72 hour
  in single ascending dose cohort
AUCtau: Area under the plasma concentration-time curve from time 0 to tau(dosing interval) | Day1 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour, Day 4, 7, 10, 13 0 hour (pre dose), Day 15 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in multiple ascending dose cohort
T1/2: Elimination half-life | 0 hour (pre-dose), 0.25 hour, 0.5 hour, 0.75 hour, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour, 10 hour, 12hour, 24 hour, 36 hour, 48 hour, 72 hour
  in single ascending dose cohort
T1/2: Elimination half-life | Day1 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour, Day 4, 7, 10, 13 0 hour (pre dose), Day 15 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in multiple ascending dose cohort
concentration of serum glucose | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in single ascending dose cohort
concentration of serum glucose | Day 1 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour, Day 4, 7, 10, 13 pre dose, Day 15 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in multiple ascending dose cohort
concentration of insulin | Day -1 pre dose, 0.5, 1, 1.5, 2, 3, 4 hour, Day 15 pre dose, 0.5, 1, 1.5, 2, 3, 4 hour
  in multiple ascending dose cohort
Changes from baseline for Body weight in kilograms | Day -1 0 hour, Day 15 0 hour
  in multiple ascending dose cohort
Changes from baseline for HbA1C in percent | Day -1 0 hour, Day 15 0 hour
  in multiple ascending dose cohort
concentration of Urine glucose excretion | 0(pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in single ascending dose cohort
concentration of Urine glucose excretion | Day 1 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour, Day 4, 7, 10, 13 pre dose, Day 15 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hour
  in multiple ascending dose cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea